CLINICAL TRIAL: NCT07394010
Title: The Role of Cardiopulmonary Exercise Testing in People With Heart Failure With Preserved Ejection Fraction
Brief Title: Role of Cardiopulmonary Exercise Testing in People With Heart Failure With Preserved Ejection Fraction
Status: Completed | Type: Observational
Sponsor: University of Ulster (Other)
Collaborators: Ulster Hospital, Northern Ireland (Unknown)
Responsible Party: Sponsor
Other Study IDs: FCNUR-23-066; 23/NI/0167 (Other: Regional Ethical Committee Northern Ireland); IRAS Project ID:32821 (Other: Health Research Agency, UK)
Record Dates: First submitted 2026-01-21; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFPEF)
Keywords: Cardiopulmonary Exercise Testing; CPET; HFpEF; Heart Failure with Preserved Ejection Fraction
MeSH Terms: interventions — Exercise Test; Clostridium perfringens epsilon-toxin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patents referred to Cardiology Department with a clinical suspicion of HFpEF: Males and Females Age range: 18 to 80 Ejection fraction >50% on the latest Echocardiography No Hospital admission in the past 6 months No pregnant No absolute contraindication for conducting an exercise test.
  Interventions: Other: Cardiopulmonary Exercise Test

INTERVENTIONS:
Other: Cardiopulmonary Exercise Test — It is the gold standard for assessing cardiorespiratory fitness. It assesses the combined functional capacity of the multiple systems of the body.
  Other Names: CPET

SUMMARY:
Heart failure affects 1-2% of the adult population. Up to half of these patients have apparently normal heart pumping function, known as heart failure with preserved ejection fraction (HFpEF). Because HFpEF typically occurs in elderly patients with multiple comorbidities, many different mechanisms could drive symptoms and life expectancy, and it has been difficult to find effective treatments that work for all. Symptoms of HFpEF occur during exertion. The current scoring system for the diagnosis of HFpEF is not able to identify the majority of people and the majority of people remain in the zone of diagnostic uncertainty; there is no definite follow-up strategy, thus people do not receive appropriate treatment. Also, the medications, prehabilitation, and rehabilitation services are not personalised.

To cater to these gaps in clinical practice, this study was set up to use Cardiopulmonary exercise testing (CPET) to understand the complexity of this disease. The investigators plan to recruit patients with clinical suspicion of HFpEF, referred to the Cardiology Department at Ulster Hospital, Belfast, UK. After screening the medical records of patients based on the inclusion and exclusion criteria, the investigators recruited 40 patients to undergo a cardiopulmonary exercise test. CPET parameters related to the heart, lungs and muscles were recorded in real time, as the patient exercised on the bike to maximal effort.

The CPET data were then analysed to answer the above-mentioned clinical gaps. To disseminate the findings, the investigators plan to present the results at scientific, clinical, and patient group meetings and publish the findings in medical journals, to reach a wide array of healthcare professionals and policymakers.

DETAILED DESCRIPTION:
The Patient Public Involvement (PPi) panel was formed. To recruit PPi members for the present study, a poster was developed to invite people to join the PPi group. It was posted on social media and shared with local community groups and as a result, a four-member PPi panel was formed during the study development phase. The PPi group consisted of 3 males and 1 female. All four PPi group members had been diagnosed and living with heart failure for over 10 years. The PPi group members gave their valuable input:

* To enhance the acceptability and feasibility of the study by helping to optimize the testing protocol for patient comfort and safety.
* To ensure that patient information materials and consent processes were clear, patient-friendly and understandable.
* To improve recruitment by identifying potential barriers by providing strategies such as waving off hospital parking ticket fee.
* To direct the objectives and interpretation of research findings in a way that is meaningful to the patients and the public.

The study was conducted in compliance with the data protection regulations and ethical research practices. Measures were taken to safeguard participant information and research data. All data collection, storage and processing adhered to the UK General Data Protection Regulation (GDPR) principles thus maintaining data integrity and confidentiality. Personal identifiable patient data was anonymised by allocating each patient a study number/ID. A master file was created and stored separately that linked the patient files with the anonymised data sheets. Anonymised data was used for SPSS analysis and for any results presentation purposes.

As part of the biological Quality Control, a healthy subject volunteered to undergo cardiopulmonary testing at 2 separate times (start and end) during the data collection.

A multi-stage consent approach was practiced. Patients were contacted via phone call by the cardiology registrar (direct care team), briefly explaining the study details and seeking interest and verbal consent to post out the participant information sheet (PIS). The contact details of those patients were passed on to the external research team (PhD researcher). Days later, those patients were contacted again via phone call by the clinical researcher explaining the study in detail, answering queries and asking their verbal consent to send out a formal appointment letter for a mutually agreed date and time.

On the day of testing, formal written informed consent was obtained that included signing both the University consent form and the Hospital consent form. It was done after the patients received clear information about the procedure, benefits, and risks.

Cardiopulmonary Exercise Test Protocol:

The CPET involved four phases: the resting phase, the warm-up phase, the incremental exercise phase, and the recovery phase.

Rest Phase Lasting between 2-3 minutes, the purpose of the resting phase was to allow patients to familiarize themselves with the equipment and for recording resting measurements (Radtke et al. 2019). Resting state values for VO2, respiratory exchange ratio (RER), and minute ventilation (VE) and heart rate were recorded and assessed for any abnormal values. Resting BP was recorded and 12-Lead ECG tracings shown on the screen were checked for any abnormalities. The printed Borg-10 scale was shown to the patients to point out their baseline scores for leg fatigue and breathlessness. Once all the checks were found to be within their desired range, the test progressed to the warm-up phase.

Warm-up/Unloaded Phase During the warm-up phase, lasting 2 minutes, the patients were asked to pedal on the cycle ergometer at zero workload (unloaded) with a pedaling cadence between 55 and 70 revolutions per minute (rpm). This was to build up a metabolic demand on the body systems to move the limbs used for exercise only. It was observed that the heart rate and breathing rate due to anxiety lowered and stabilized once the patient began to cycle to match the metabolic requirement. One minute into the warm-up phase, blood pressure was recorded. After 2 minutes, the test progressed onto the incremental exercise phase automatically.

Incremental/Loaded Exercise Phase Lasting 10 ± 2 minutes, this phase involved a gradual (ramped) increase in exercise intensity. The workload (resistance required to turn the flywheel) increased at a pre-defined/calculated rate for the duration that the patient was able to continue cycling. The patients were motivated to keep cycling against the workload till they reached their maximal exhaustion while keeping the cadence above 55 rpm at all times. During the phase, CPET parameters were recorded and displayed on the screen in real time. Additional parameters were recorded at multiple checkpoints pre-set in the protocol. This included blood pressure recordings at 2 minutes interval at the initial segment of the phase followed 1 minute interval once the respiratory exchange ratio was seen to cross 1.0 mark. The perceived exertion assessed via the Borg-10 scale was recorded at 4 minutes into the test and as close to maximal exhaustion as possible. The test was switched to the recovery phase at the point where the patients raised their hand, signalling that they were maximally exhausted.

Recovery The recovery phase lasted for 3-5 minutes, during which the load on the bike was reduced to zero watts and variables were continually monitored to measure the patients' ability to recover from the exercise protocol. Serial BP readings were taken at every 2-minute intervals. During the recovery period, the patients continued to cycle at the same cadence to maintain the blood flow in the lower limbs and remove by-products of exercise (e.g. lactate build-up) The test was terminated once VO2 had returned to 50% of the peak values or the heart rate and systolic BP return to within the 20 beats/min and 20mm Hg of the pretest resting values respectively. Once the recovery data was collected, the patients were asked to warm down to a state of complete rest.

Continuous Monitoring throughout CPET Continuous monitoring of all the CPET variables was done throughout the exercise test by the CPET lead (PhD researcher). Particularly during the incremental workload phase, the rising VO2 , VCO2, VE and HR curves and BP readings were monitored to ensure that the test was being conducted both efficiently and safely.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Age range between 18 - 80 years
* Clinical suspicion of Heart failure with preserved ejection fraction
* Ejection Fraction of ≥50% on the most recent Echocardiogram
* Able to understand the performance of an exercise test and the ability to provide consent
* Ability to undertake leg exercise without any impediment

Exclusion Criteria:

* • Hospital admission in the past 6 months

  * Unable to understand the performance of an exercise test
  * Unable to provide informed consent
  * Female subjects who are knowingly pregnant or believe they may be pregnant
  * Having an impediment preventing them from performing cycle ergometry
  * Contra-indication of CPET: acute myocardial infarction, unstable angina, uncontrolled arrhythmias, moderate or severe valvular disease, High-degree atrioventricular block, acute infection, acute endocarditis, myocarditis, uncontrolled asthma, and history of syncope.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients registered with the South Eastern Health and Social Trust (NHS), Northern Ireland, UK.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Maximum Oxygen Consumption at peak exercise (VO2peak) | CPET testing day. VO2peak is recorded as the oxygen consumption value measured by the gas sensor at the peak of exercise, i.e., seconds before maximal exhaustion.
  Measure of exercise capacity.

SECONDARY OUTCOMES:
First Ventilatory Threshold | CPET testing day. Measured during the initial 3 minutes of the incremental test phase.
  Exercise intensity at which lactate levels start to rise exponentially
Heart Rate | Baseline, every 2 minutes interval, and at peak exercise near maximal exhaustion.
  The rate at which the heart beats. Measured in beats per minute throughout the exercise test.
Blood Pressure | Every 3-minute interval during the exercise test.
  Mean blood pressure in the main artery during pumping and relaxation phase of the heart

CONTACTS AND LOCATIONS:
Overall Officials: Chris Bleakley, PhD, Study Director — Ulster University, Belfast, UK; George Kernohan, PhD, Study Director — Ulster University, Belfast, UK; Peter McKavanagh, MD, PhD, Study Director — Ulster Hospital
Locations (1):
- Ulster University and Ulster Hospital, Belfast, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol
Time Frame: From March 2026 onwards
Access Criteria: Freely available online for anyone to access
URL: https://pure.ulster.ac.uk/en/persons/saqib-javaid/

REFERENCES:
- See also: Cardiopulmonary exercise testing in heart failure with preserved ejection fraction: a game-changer for patients. — https://bmjopenrespres.bmj.com/content/12/Suppl_1/A31.1

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2026-01-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT07394010/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT07394010/ICF_001.pdf